CLINICAL TRIAL: NCT00007774
Title: CSP #451 - The Clinical and Economic Impact of Olanzapine in the Treatment of Schizophrenia
Brief Title: To Determine if Olanzapine is More Cost Effective Than Haloperidol for the Treatment of Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Rosenheck, Robert - Study Chair, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Masking: Double
Other Study IDs: 451
Record Dates: First submitted 2000-12-29; First posted 2001-01-01 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Schizoaffective Disorder; Schizophrenia
Keywords: Olanzapine, haloperidol, schizophrenia, schisoaffe
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Haloperidol; Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Olanzapine
  Interventions: Drug: Olanzapine
- 2 (Active Comparator): Haloperidol
  Interventions: Drug: Haloperidol

INTERVENTIONS:
Drug: Haloperidol
  Arms: 2
Drug: Olanzapine
  Arms: 1

SUMMARY:
Although currently marketed antipsychotic drugs are useful in the treatment of schizophrenia, efficacy and safety profiles need to be improved. Forty to eighty percent of patients either fail to respond or only partially respond to conventional antipsychotic agents. Secondary symptoms may be unimproved even in patients who respond to treatment. A variety of adverse events occur in patients receiving currently available agents. The severity of these events contributes to the poor compliance that is observed in this patient population. Olanzapine is a novel antipsychotic agent with a reduced incidence of extrapyramidal symptoms. Other side effects are minimal.

DETAILED DESCRIPTION:
Primary Hypothesis: To determine if olanzapine is more cost effective than haloperidol for the treatment of schizophrenia.

Secondary Hypothesis: Secondary objectives include evaluation of clinical efficacy, safety, social and vocational functioning, family burden, compliance and satisfaction for olanzapine relative to haloperidol.

Intervention: Olanzapine (5 mg to 20 mg/day), haloperidol (5 mg to 20 mg/day).

Primary Outcomes: Total inpatient hospital care costs are the primary outcome. Other major outcomes are total social costs (cost of VA health care, non-VA services and other specified social costs), efficacy measures (PANNS, BPRS, CGI Severity, and neurocognitive battery scores) and safety measures (adverse events, ECG?s).

Study Abstract: Although currently marketed antipsychotic drugs are useful in the treatment of schizophrenia, efficacy and safety profiles need to be improved. Forty to eighty percent of patients either fail to respond or only partially respond to conventional antipsychotic agents. Secondary symptoms may be unimproved even in patients who respond to treatment. A variety of adverse events occur in patients receiving currently available agents. The severity of these events contributes to the poor compliance that is observed in this patient population. Olanzapine is a novel antipsychotic agent with a reduced incidence of extrapyramidal symptoms. Other side effects are minimal.

Approximately 327 patients with schizophrenia or schizoaffective disorder were randomly assigned to one of two treatment groups. One treatment group was prescribed olanzapine with daily dosage ranging from 5 mg/day to 20 mg/day. The other treatment group was prescribed haloperidol with daily dosage also ranging from 5 mg/day to 20 mg/day. A semi-structured psychosocial case management treatment program is provided for all study patients. Patients were recruited from 18 VA medical centers over a 24-month period and were followed for one year. 18 patients were enrolled at one site that had its research program terminated during the study. Because of questions regarding the circumstances that led to the termination, these 18 patients will not be included in study analyses. The major objective of the study is to determine if olanzapine is more cost effective than haloperidol. Secondary objectives include evaluation of clinical efficacy, safety, social and vocational functioning, family burden, compliance and satisfaction for olanzapine relative to haloperidol.

MANUSCRIPT: Primary manuscript published in JAMA, November 2003.

ELIGIBILITY:
Inclusion Criteria:

Patients with schizophrenia or schizoaffective disorder.

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 1998-03; Primary Completion 2001-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Rosenheck, AB MD, Study Chair — VA Connecticut Health Care System (West Haven)
Locations (18):
- United States (18):
  - VA Medical Center, Tuscaloosa, Tuscaloosa, Alabama
  - VA Palo Alto Health Care System, Palo Alto, California
  - VA Connecticut Health Care System (West Haven), West Haven, Connecticut
  - VA Medical Center, Bay Pines, Bay Pines, Florida
  - VA Medical Center, Miami, Miami, Florida
  - VA Medical Center, Augusta, Augusta, Georgia
  - Richard Roudebush VA Medical Center, Indianapolis, Indianapolis, Indiana
  - VA Maryland HCS, Perry Point Division, Perry Point, Maryland
  - Edith Nourse Rogers Memorial Veterans Hospital, Bedford, Bedford, Massachusetts
  - John D. Dingell VA Medical Center, Detroit, Detroit, Michigan
  - VA New Jersey Health Care System, East Orange, East Orange, New Jersey
  - New Mexico VA Health Care System, Albuquerque, Albuquerque, New Mexico
  - Franklin Delano Roosevelt Campus, VA Hudson Valley HCS, Montrose, New York
  - New York Harbor HCS, New York, New York
  - VA Medical Center, Durham, Durham, North Carolina
  - VA Medical Center, Cleveland, Cleveland, Ohio
  - VA Medical Center, Philadelphia, Philadelphia, Pennsylvania
  - VA Pittsburgh Health Care System, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Perlick DA, Rosenheck RA, Kaczynski R, Bingham S, Collins J. Association of symptomatology and cognitive deficits to functional capacity in schizophrenia. Schizophr Res. 2008 Feb;99(1-3):192-9. doi: 10.1016/j.schres.2007.08.009. Epub 2007 Sep 12. PMID 17851042
- [Result] Rosenheck R, Perlick D, Bingham S, Liu-Mares W, Collins J, Warren S, Leslie D, Allan E, Campbell EC, Caroff S, Corwin J, Davis L, Douyon R, Dunn L, Evans D, Frecska E, Grabowski J, Graeber D, Herz L, Kwon K, Lawson W, Mena F, Sheikh J, Smelson D, Smith-Gamble V; Department of Veterans Affairs Cooperative Study Group on the Cost-Effectiveness of Olanzapine. Effectiveness and cost of olanzapine and haloperidol in the treatment of schizophrenia: a randomized controlled trial. JAMA. 2003 Nov 26;290(20):2693-702. doi: 10.1001/jama.290.20.2693. PMID 14645311